CLINICAL TRIAL: NCT04020757
Title: H+ Mobilization With Dialysate Bicarbonate Variation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Biochemical measurement techniques were deemed insufficient to continue research
Sponsor: Tufts Medical Center (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 13296
Record Dates: First submitted 2019-06-04; First posted 2019-07-16 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bicarb Variation (Other): Variation in dialysis bicarbonate, lowered to 30 mEq/L for week 2 of 3
  Interventions: Device: variation in dialysis bicarbonate; Dietary Supplement: Zone Perfect bar

INTERVENTIONS:
Device: variation in dialysis bicarbonate — 35 mEq/L dialysate bicarbonate for one week, followed by 30 mEq/L for one week, followed by 35mEq/L for one week with nutritional supplement during dialysis
Dietary Supplement: Zone Perfect bar — 16g protein supplement given during first 30 mins of dialysis on last testing day

SUMMARY:
The aims of the proposed studies are first to delineate the physiological response of End Stage Kidney Disease (ESKD) patients to exposure to a bath [HCO3-] of 35 mEq/L and an [acetate] of 4 mEq/L, and second, to determine whether reducing bath [HCO3-] will have the expected effect of decreasing or abolishing stimulation of organic acid production. A secondary endpoint will be whether the patients tolerate such a reduction and its impact on pre-dialysis blood [HCO3-]. If the outcome is positive in both regards, future studies will measure well-being and outcomes with reduced bath [HCO3-].

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years or older,
2. Have been on dialysis for at least 1 year,
3. Be stable on treatment (i.e., without frequent changes in their dialysis prescription, or recent hospitalizations),
4. Be reasonably nourished (serum albumin > 3.5 g/dl and not currently receiving oral nutritional supplement through DCI).
5. Self-reported urine output of <200 cc/day
6. Functioning arteriovenous fistulas or grafts for dialysis access
7. Currently dialyzing at a dialysate [HCO3-] of 33-37 mEq/L.

Exclusion Criteria:

1. Pregnancy,
2. Acute illnesses of any kind,
3. Hospitalization in the prior 3 months (except for vascular access related),
4. Significant congestive heart failure, liver or lung failure.
5. Pre-dialysis blood [HCO3-] <19 mEq/L) (to reduce the risk of metabolic acidosis )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Lactate levels | through study completion, a period of 3 weeks
  7 tests conducted through the dialysis treatment after the long interdialytic interval
H+ mobilization | through study completion, a period of 3 weeks
  7 tests conducted through the dialysis treatment after the long interdialytic interval

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States